CLINICAL TRIAL: NCT05654571
Title: Evaluation of the Relationship Between Weight Loss and Breast Cancer After Laparoscopic Sleeve Gastrectomy Surgery
Brief Title: Weight Loss and Breast Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ANIL ERGIN, Uzman Doktor, Fatih Sultan Mehmet Training and Research Hospital
Other Study IDs: ANILERGİNN
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Breast Cancer; Obesity, Morbid
Keywords: breast cancer; obesity; laparoscopic sleeve gastrectomy; wight loss; mammography
MeSH Terms: conditions — Breast Neoplasms; Obesity, Morbid; Obesity | interventions — Mammography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- significant weight loss+ breast cancer: The group that lost significant weight after laparoscopic sleeve gastrectomy and was diagnosed with breast cancer
  Interventions: Diagnostic Test: mammography
- regain+breast cancer: The group who lost significant weight after laparoscopic sleeve gastrectomy and regained it afterwards, or who could not lose weight and were diagnosed with breast cancer
  Interventions: Diagnostic Test: mammography

INTERVENTIONS:
Diagnostic Test: mammography — All patients are checked for mammography every year after surgery.

SUMMARY:
Obesity is an important risk factor for postmenopausal breast cancer. A large meta-analysis concluded that obesity is associated with a 20% to 40% increased risk for receptor-positive postmenopausal breast cancer. The International Agency for Research on Cancer working group on obesity and cancer risk drew similar conclusions. Obesity seems to have the opposite effect among premenopausal women, with most studies suggesting that higher BMI is associated with a reduced risk of premenopausal breast cancer.

Determining whether deliberate weight loss is associated with a reduced risk of breast cancer is difficult in part because sustained weight loss is difficult to achieve and few studies have sufficient statistical power to address this question. Bariatric surgery is one of the few weight loss interventions in which significant weight loss is maintained. A limited number of previous studies have suggested a reduced risk of cancer following bariatric surgery. Recently, it showed that bariatric surgery is associated with a lower risk of several types of cancer, including an approximately 40 % reduction in the risk of postmenopausal breast cancer. However, whether bariatric surgery affects breast cancer risk in premenopausal women and whether this association is altered by estrogen receptor (ER) status has not been addressed.

The aim of this study is to examine the relationship between weight loss after laparoscopic sleeve gastrectomy (LSG) and breast cancer.

DETAILED DESCRIPTION:
In this study, 300 female patients who underwent laparoscopic sleeve gastrectomy due to morbid obesity in Fatih Sultan Mehmet Training and Research Hospital General Surgery Clinic will be included. The number of samples was calculated by performing impact power analysis.

Mamagrophy is recommended for all women over the age of 40 as part of the routine cancer screening program in our country. For this reason, it is assumed that female patients over the age of 40 who have undergone LSG operation have undergone mammography as of 2022. For this reason, the data of these patients will be examined by scanning from the hospital system. Patients who have undergone mammography examination at least 3 years after the LSG operation will be included in the study. The mammograms of the patients who underwent mammography in January 2015 and later will be evaluated. The final diagnosis of breast cancer will be made with the pathology result in patients with suspicious appearance on mamagrophy.

If there is a malignancy detected as a result of the examinations, its size and pathology will be recorded. Patients' age, gender, and total weight loss will be recorded.

In this retrospective study, we aimed to determine the incidence of breast cancer in patients who had undergone LSG surgery and also to determine whether there was a change in breast cancer compared to weight loss.

The patient inclusion criteria are as follows:

* 40 years and older (age as of 2022, not the age of operation)
* LSG was applied in our clinic due to morbid obesity.
* Patients whose mamagrofi images are available in the hospital system

The patient exclusion criteria are as follows:

* Patients who underwent abdominal surgery again after LSG
* Patients whose mamagrophy image is not in the system
* Patients with suspicious findings as a result of mammography and who did not undergo additional imaging or biopsy
* Patients out of follow-up after the operation

ELIGIBILITY:
Inclusion Criteria:

* 40 years and older (age as of 2022, not the age of operation)
* LSG was applied in our clinic due to morbid obesity.
* Patients whose mamagrofi images are available in the hospital system

Exclusion Criteria:

* Patients who underwent abdominal surgery again after LSG
* Patients whose mamagrophy image is not in the system
* Patients with suspicious findings as a result of mammography and who did not undergo additional imaging or biopsy
* Patients out of follow-up after the operation

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Since the incidence of breast cancer was investigated in the study and the incidence of breast cancer in women is much higher than in men, only female patients will be included. Since all patients included in the study would undergo mammography, female patients over the age of 40 were included in the study.
Study Population: female patients over 40 years of age
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-12-15 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
breast cancer incidence after laparoscopic sleeve gastrectomy | 5 year
  Comparison of breast cancer incidence in those who lost weight after laparoscopic sleeve gastrectomy and those who did not.

SECONDARY OUTCOMES:
breast cancer incidance | 5 year
  Comparison of breast cancer incidence in those who lose weight after laparoscopic sleeve gastrectomy with the normal population

CONTACTS AND LOCATIONS:
Locations (1):
- Fatih Sultan Mehmet Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
If there is a request for the sharing of data, it will be shared.